CLINICAL TRIAL: NCT00096057
Title: An Open Label Phase I Study of Humanized Human Milk Fat Globule-1 (huHMFG1) Antibody in Patients With Locally Advanced or Metastatic Breast Cancer (TOPCAT)
Brief Title: Monoclonal Antibody HuHMFG1 in Treating Women With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: ROCHE-NP17787; UCLA-0402065-01; CDR0000391212 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — epitumomab

INTERVENTIONS:
Biological: monoclonal antibody HuHMFG1

SUMMARY:
RATIONALE: Monoclonal antibodies such as HuHMFG1 can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: This phase I trial is studying the side effects and best dose of monoclonal antibody HuHMFG1 in treating women with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of monoclonal antibody HuHMFG1 in women with locally advanced or metastatic breast cancer.
* Determine a safe recommended dose and schedule of this drug in these patients.
* Determine the pharmacokinetic profile, in the absence of any other chemotherapy or endocrine agent, of this drug in these patients.
* Determine the antitumor activity of this drug in these patients.
* Determine time to progression in patients treated with this drug.
* Assess immunological markers (e.g., granzyme B, gamma interferon, and C1Q) for determining response to this drug in these patients.
* Assess markers of immunogenicity (e.g., human anti-human antibody) of this drug in these patients.
* Assess tumor markers (e.g., CA15.3 and CEA) in patients treated with this drug.
* Correlate, preliminarily, soluble HMFG1 antigen levels with pharmacokinetic data for this drug in these patients.

OUTLINE: This is an open-label, non-randomized, dose-escalation study.

Patients in cohorts 1 and 2 receive monoclonal antibody HuHMFG1 IV over 1-3 hours once every 21 days for doses 1 and 2. All subsequent dose intervals are based on individual half-life value of the drug, to be within 3 days of the estimated half-life in multiples of 7 days. Patients in cohorts 3 and 4 receive monoclonal antibody HuHMFG1 at the dosing interval determined in the first 2 cohorts. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of monoclonal antibody HuHMFG1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

All patients are followed at 4 weeks and then every 6 weeks for 6 months. Patients with an antitumor response or stable disease are followed every 12 weeks until disease progression or initiation of another antitumor treatment.

PROJECTED ACCRUAL: A total of 6-24 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Locally advanced or metastatic disease
  * No inflammatory breast cancer
* Measurable (RECIST) or evaluable disease (e.g., cytologically or radiologically detectable disease that does not fulfill RECIST criteria)
* Failed prior OR not a candidate for OR refused anthracycline- and taxane-containing chemotherapy
* Patients whose tumor overexpresses HER-2 must have failed prior trastuzumab (Herceptin®)
* No known CNS metastases
* No metastases accessible to complete surgical resection
* Unstained slides cut from formalin-fixed and paraffin-embedded tumor blocks available

  * Appropriate tumor block also acceptable
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* WHO 0-1

Life expectancy

* At least 4 months

Hematopoietic

* Hemoglobin ≥ 10 g/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* WBC ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* ALT or AST ≤ 2.5 times upper limit of normal (ULN) (< 5 times ULN in patients with liver metastases) OR
* Alkaline phosphatase ≤ 2.5 times ULN (< 5 times ULN in patients with liver metastases)

  * Any degree of elevated alkaline phosphatase allowed provided it is due to bone metastases

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance > 60 mL/min
* Uric acid < 1.25 times ULN (for patients with hyperuricemia only)
* Calcium (corrected for serum albumin) < 11.5 mg/dL (for patients with hypercalcemia only)

Cardiovascular

* LVEF ≥ 45% by MUGA or echocardiogram within the past 4 weeks

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or cervical intra-epithelial neoplasia
* No other uncontrolled illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* Prior biological therapy allowed
* More than 2 weeks since prior blood transfusions or growth factors to aid hematological recovery
* No other concurrent antitumor immunotherapy

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior cytotoxic chemotherapy
* No more than 3 prior chemotherapy regimens, including adjuvant/neoadjuvant therapy
* No concurrent antitumor chemotherapy

Endocrine therapy

* Prior hormonal therapy allowed
* No concurrent corticosteroids except as physiologic replacement and/or for acute short-term treatment of, or prophylaxis against, infusion reactions
* No concurrent antitumor hormonal therapy

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy (except for palliative radiotherapy)
* No concurrent antitumor radiotherapy, except for palliation to non-study lesions

  * Irradiated area should be as small as possible and involve ≤ 10% of the bone marrow in any given 4-week period

Surgery

* More than 4 weeks since prior major surgery

Other

* More than 30 days since prior investigational agents
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2004-05; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Pegram, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Derived] Pegram MD, Borges VF, Ibrahim N, Fuloria J, Shapiro C, Perez S, Wang K, Schaedli Stark F, Courtenay Luck N. Phase I dose escalation pharmacokinetic assessment of intravenous humanized anti-MUC1 antibody AS1402 in patients with advanced breast cancer. Breast Cancer Res. 2009;11(5):R73. doi: 10.1186/bcr2409. PMID 19811637